CLINICAL TRIAL: NCT04687384
Title: Systemic and Peritoneal Inflammatory Response In Robotic-assisted And Laparoscopic Surgery for Colon Cancer (SIRIRALS-trial): a Randomized Controlled Trial
Brief Title: Systemic and Peritoneal Inflammatory Response In Robotic-assisted And Laparoscopic Surgery for Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 75709
Record Dates: First submitted 2020-11-27; First posted 2020-12-29 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Colonic Neoplasms; Colon Cancer; Systemic Inflammatory Response Syndrome; Inflammation; Robotic Surgical Procedures; Laparoscopy; Peritoneal Inflammation
Keywords: Systemic inflammatory response; Colonic neoplasm; Robotic assisted surgery; Laparoscopy
MeSH Terms: conditions — Colonic Neoplasms; Systemic Inflammatory Response Syndrome; Inflammation; Peritonitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic-assisted surgery (Experimental): Patients undergoing robotic-assisted colectomy for colonic neoplasm
  Interventions: Procedure: Robotic-assisted colectomy
- Laparoscopy (Active Comparator): Patients undergoing conventional laparoscopic colectomy for colonic neoplasm
  Interventions: Procedure: Conventional laparoscopic colectomy

INTERVENTIONS:
Procedure: Robotic-assisted colectomy — Robotic-assisted colectomy performed by usage of da Vinci Xi robotic technology
  Arms: Robotic-assisted surgery
Procedure: Conventional laparoscopic colectomy — Conventional laparoscopic colectomy
  Arms: Laparoscopy

SUMMARY:
The current hypothesis is that robotic-assisted surgery results in a reduced systemic and peritoneal inflammatory response (SIRS) compared to laparoscopic surgery in the treatment of colon cancer. The purpose is to evaluate differences in the peritoneal and systemic inflammatory response in robot-assisted and laparoscopic surgery of patients undergoing resection for colon cancer in a randomized, blinded controlled trial.

ELIGIBILITY:
Inclusion criteria

* Elective robotic-assisted or laparoscopic surgery for right-sided, left-sided and sigmoid colon cancer
* Aged ≥ 18
* ASA-score ≤ 3
* Tumor-stage (Tx-T4a)
* Endoscopic suspected colon cancer
* Histological verified adenocarcinoma, signet ring cell carcinoma, undifferentiated cancer, medullary carcinoma, or another malignant tumor type originating from colon
* Patients must give informed written consent
* Patients must be able to understand Danish language

Exclusion criteria

* Carcinoma of the transverse colon or synchronous colorectal cancer
* Previous history of colon cancer
* Previous open major abdominal surgery with exception of open appendectomy and cholecystectomy.
* Metastatic disease
* Pregnancy
* History of psychiatric or addictive disorder that would prevent the patient from participating in the trial
* Emergency colon surgery
* Co-existing inflammatory bowel disease
* Co-existing immunological disease that requiring ingestion of systemic immunomodulatory drugs (DMARD - disease modifying anti-rheumatic drugs), corticosteroids and biologic disease-modifying anti-rheumatic drugs.
* Daily consumption of NSAID drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in levels of systemic inflammatory response expressed by CRP and IL-6 in serum between the two groups | Baseline and postoperative (day 1-3)
  CRP (mg/L), IL-6 (pg/mL)

SECONDARY OUTCOMES:
Changes in levels of systemic inflammation in serum between the two groups | Baseline and postoperative (day 1-3)
  The cytokine levels are expressed by: Eotaxin, Eotaxin-3, GM-CSF, IFN-γ, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-7, IL-8, IL-8 (HA), IL-10, IL-12/IL-23p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, TARC, TNF-α, TNF-β, VEGF-A and IL-1RA. All cytokines are measured in pg/mL
Differences in number of patients with postoperative surgical and medical complications (30 days) according to Clavien-Dindo classification and Comprehensive Complication Index (CCI) | 30 days
  Number of complications obtained from medical records
Differences in intraoperative blood loss | 1 day
  Measured in mL
Conversion rate to open surgery | 1 day
  Number of conversions to open surgery
Length of surgery (total anesthesia time) | 1 day
  Measured in minutes
Length of surgery (total surgical time) | 1 day
  Measured in minutes
Lymph node yield | 14 days
  Pathological examination of lymph nodes
Length of hospital stay | 14 days
  Measured in days
Postoperative pain | Baseline and postoperative (day 1-3 and 14)
  Measured by VAS-scale
Time to first flatus | Postoperative (day 1-3)
  Measured in hours
Time to first bowel movement | Postoperative (day 1-3)
  Measured in hours

OTHER OUTCOMES:
Levels of peritoneal inflammatory response in peritoneal fluid | Postoperative (day 1-3)
  Levels of cytokines are expressed by: Eotaxin, Eotaxin-3, GM-CSF, IFN-γ, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, IL-12/IL-23p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, TARC, TNF-α, TNF-β, VEGF-A as well as IL-1RA and CRP. All cytokines are measured in pg/mL, CRP measured in mg/L
Patient reported health related quality of recovery (QoR-15) | Baseline and postoperative (day 1-3 and 14)
  Recovery is measured according to quality of recovery 15 score (QoR-15). The score ranges from 0-150. A high score indicates a good recovery.
Mortality | 30 days
  Number of mortality obtained from medical charts
Heart rate variability | Postoperative (day 1-3)
  The heart rate will continuously recorded by ECG intra- and postoperatively
Whole blood gene expression profiling | Baseline and postoperative (day 1-3)
  Gene mRNA transcript analysis
Time to local cancer recurrence or metastatic spread | 3 years postoperatively
  The two surgical methods will be compared in order to obtain any differences in the local or metastatic cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Pedja Cuk, MD, Principal Investigator — Surgical Department, Hospital of Southern Jutland, Denmark
Locations (1):
- Hospital of Southern Denmark, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuk P, Tiskus M, Moller S, Lambertsen KL, Backer Mogensen C, Festersen Nielsen M, Helligso P, Gogenur I, Bremholm Ellebaek M. Surgical stress response in robot-assisted versus laparoscopic surgery for colon cancer (SIRIRALS): randomized clinical trial. Br J Surg. 2024 Mar 2;111(3):znae049. doi: 10.1093/bjs/znae049. PMID 38445434
- [Derived] Cuk P, Pedersen AK, Lambertsen KL, Mogensen CB, Nielsen MF, Helligso P, Gogenur I, Ellebaek MB. Systemic inflammatory response in robot-assisted and laparoscopic surgery for colon cancer (SIRIRALS): study protocol of a randomized controlled trial. BMC Surg. 2021 Oct 11;21(1):363. doi: 10.1186/s12893-021-01355-4. PMID 34635066